CLINICAL TRIAL: NCT01457040
Title: A Prospective Study of Intensified Conditioning Regimen With High-Dose-Etoposide for Allogeneic Hematopoietic Stem Cell Transplantation for Adult Acute Lymphoblastic Leukemia in China
Brief Title: Intensified Conditioning Regimen With High-Dose-Etoposide for Allo-HSCT for Adult Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Hongsheng Zhou, Professor, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDE-ALL-2011
Record Dates: First submitted 2011-10-11; First posted 2011-10-21 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2015-10

CONDITIONS: Acute Lymphoblastic Leukemia; Stem Cell Transplantation, Hematopoietic
Keywords: Acute Lymphoblastic leukemia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complete Remission (CR) (Experimental): CR Cohort: high-risk ALL in CR and standard-risk ALL in the status of ≥CR2
  Interventions: Drug: TBI+CY+VP-16
- Non-Remission (NR) (Experimental): NR Cohort: ALL in non-remission
  Interventions: Drug: FA+TBI+CY+VP-16

INTERVENTIONS:
Drug: TBI+CY+VP-16 — CR Cohort will receive conditioning regimen of TBI+CY+VP-16: TBI: 4.5Gy/d, -5d, -4d; CY: 60mg/kg/d, -3d, -2d; VP-16: 15mg/kg/d, -3d, -2d
  Arms: Complete Remission (CR)
Drug: FA+TBI+CY+VP-16 — NR Cohort will receive conditioning regimen of FA+TBI+CY+VP-16: Flu: 35mg/m2/d: -10~-6d; AraC: 1g/m2/d, -10d~-6d; TBI: 4.5Gy/d, -5d,-4d; CY:60mg/kg/d, -3d, -2d; VP-16: 15mg/kg, -3d, -2d
  Arms: Non-Remission (NR)

SUMMARY:
Evolving paradigms in the treatment of adult ALL include the application of intense pediatric regimens to the treatment of adolescents and young adults (AYA) and the optimization of allogeneic hematopoietic stem cell transplantation (allo-HSCT) in the cure of patients. The Cancer and Leukemia Group B (CALGB) and the Children's Cancer Group (CCG) first asked whether AYA between the ages of 16 and 20 fared differently whether they were treated on pediatric protocols. The results of this study demonstrated that although the complete remission rates were identical for the AYAs treated on the CALGB and CCG trials, the AYAs had a 63% event-free survival (EFS) and 67% OS at 7 years on the CCG trials compared with 34% and 46%, respectively, on the CALGB trials.

High relapse and transplantation-related-mortality still remains great challenge for HSCT of adult ALL, which both range between 25% and 30%. Recently, risk-adapted indication and optimization of conditioning regimen are highlighted, which aiming to reduce TRM and relapse rate, respectively.City of Hope National Medical Center studied the substitution of etoposide (VP-16) for CY in the treatment of ALL patients receiving HCT. The result suggested that etoposide and TBI are associated with a decreased relapse rate following transplantation for ALL, compared with those receiving CY and TBI. Japanese and Germany reports pronounced the advantage of VP-16 in intensified regimen for adult ALL. On the same time, the investigators previous researches have confirmed the effect and safety of FA-intensified conditioning regimen on relapse and refractary leukemia.

Based on mentioned above, the investigators speculate that VP-16-intensified conditioning regimen could improve the outcome for adult ALL. The potential mechanism will be attributed to reduce MRD and promote GVL effect via providing enough time-window for immuno-reconstitution by high-dose preparative regimen.

DETAILED DESCRIPTION:
In the first decade of the new millennium, multiple studies have begun to change our thinking about the treatment of adults with acute lymphoblastic leukemia (ALL). In pediatric patients cure rates in the range of 80% to 90% are now attainable. While adult patients with ALL now have a 90% complete remission (CR) with modern chemotherapy, most patients will relapse, and leukemia-free survival with 3 to 7 years of follow-up in large series is only in the range of 30% to 40%. The poor outcome of chemotherapy in adults with ALL as compared to children relates to multiple factors, including poor tolerance of intensive courses of chemotherapy and a higher incidence of poor prognostic subtypes of ALL such as Philadelphia chromosome-positive ALL and a lower incidence of favorable subtypes such as the t (12; 21).

Evolving paradigms in the treatment of adult ALL include the application of intense pediatric regimens to the treatment of adolescents and young adults (AYA) and the optimization of allogeneic hematopoietic stem cell transplantation (allo-HSCT) in the cure of patients. Adult regimens are typically less intense than pediatric regimens. The Cancer and Leukemia Group B (CALGB) and the Children's Cancer Group (CCG) first asked whether AYA between the ages of 16 and 20 fared differently whether they were treated on pediatric protocols. The results of this study demonstrated that although the complete remission rates were identical for the AYAs treated on the CALGB and CCG trials, the AYAs had a 63% event-free survival (EFS) and 67% OS at 7 years on the CCG trials compared with 34% and 46%, respectively, on the CALGB trials. These results have prompted new studies where pediatric ALL regimens have been adapted to the treatment of younger adults. With short follow-up, GRAALL-2003 reports suggest EFS and OS outcomes in the range of 60%. This improved outcome was more pronounced in the standard-risk patients with a donor who had an OS at 5 years of 69%. On the same time, our previous researches have confirmed the effect and safety of FA-intensified conditioning regimen on relapse and refractary leukemia.

Based on mentioned above, we speculate that VP-16-intensified conditioning regimen could improve the outcome for adult ALL. The potential mechanism will be attributed to reduce MRD and promote GVL effect via providing enough time-window for immuno-reconstitution by high-dose preparative regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 14 years to 65 years
2. Diagnosis of High-risk acute lymphoblastic leukemia or standard-risk ALL in ≥CR2
3. Patient will receive allogeneic hematopoietic stem cell transplantation
4. The informed consent form has been signed.

Exclusion Criteria:

1. Patient with severe cardiac dysfunction with less than 50% EF
2. Patient with severe lung dysfunction
3. Patient with severe hepatic or renal dysfunction with more than 3 times the upper limit of normal range (ULN) of serum ALT or AST levels, or with more than 2 times the upper limit of normal range (ULN) of serum TBIL level or less than 40% of normal prothrombin time activity (PTA); or with more than 2 times the ULN of serum Cr
4. Patient with severe active infection
5. Patient with allergy history about suspected drug in conditioning regimen
6. Patient with other conditions considered unsuitable for the study

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Over Survival | 3 years after HSCT

SECONDARY OUTCOMES:
Leukemia-Free-Survival | 3 years after HSCT
relapse rate | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Department of Hematology, Nanfang Hospital
Locations (1):
- Department of Hematology, Nanfang Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Liu QF, Fan ZP, Zhang Y, Jiang ZJ, Wang CY, Xu D, Sun J, Xiao Y, Tan H. Sequential intensified conditioning and tapering of prophylactic immunosuppressants for graft-versus-host disease in allogeneic hematopoietic stem cell transplantation for refractory leukemia. Biol Blood Marrow Transplant. 2009 Nov;15(11):1376-85. doi: 10.1016/j.bbmt.2009.06.017. Epub 2009 Aug 19. PMID 19822296
- [Background] Ottmann OG, Pfeifer H. Management of Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL). Hematology Am Soc Hematol Educ Program. 2009:371-81. doi: 10.1182/asheducation-2009.1.371. PMID 20008223
- [Background] Laport GG, Alvarnas JC, Palmer JM, Snyder DS, Slovak ML, Cherry AM, Wong RM, Negrin RS, Blume KG, Forman SJ. Long-term remission of Philadelphia chromosome-positive acute lymphoblastic leukemia after allogeneic hematopoietic cell transplantation from matched sibling donors: a 20-year experience with the fractionated total body irradiation-etoposide regimen. Blood. 2008 Aug 1;112(3):903-9. doi: 10.1182/blood-2008-03-143115. Epub 2008 Jun 2. PMID 18519812
- [Background] Seibel NL. Treatment of acute lymphoblastic leukemia in children and adolescents: peaks and pitfalls. Hematology Am Soc Hematol Educ Program. 2008:374-80. doi: 10.1182/asheducation-2008.1.374. PMID 19074113
- [Background] Pui CH, Evans WE. Treatment of acute lymphoblastic leukemia. N Engl J Med. 2006 Jan 12;354(2):166-78. doi: 10.1056/NEJMra052603. No abstract available. PMID 16407512
- [Background] Kantarjian H, Thomas D, O'Brien S, Cortes J, Giles F, Jeha S, Bueso-Ramos CE, Pierce S, Shan J, Koller C, Beran M, Keating M, Freireich EJ. Long-term follow-up results of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone (Hyper-CVAD), a dose-intensive regimen, in adult acute lymphocytic leukemia. Cancer. 2004 Dec 15;101(12):2788-801. doi: 10.1002/cncr.20668. PMID 15481055
- [Background] Rowe JM, Buck G, Burnett AK, Chopra R, Wiernik PH, Richards SM, Lazarus HM, Franklin IM, Litzow MR, Ciobanu N, Prentice HG, Durrant J, Tallman MS, Goldstone AH; ECOG; MRC/NCRI Adult Leukemia Working Party. Induction therapy for adults with acute lymphoblastic leukemia: results of more than 1500 patients from the international ALL trial: MRC UKALL XII/ECOG E2993. Blood. 2005 Dec 1;106(12):3760-7. doi: 10.1182/blood-2005-04-1623. Epub 2005 Aug 16. PMID 16105981
- [Background] Goldstone AH, Richards SM, Lazarus HM, Tallman MS, Buck G, Fielding AK, Burnett AK, Chopra R, Wiernik PH, Foroni L, Paietta E, Litzow MR, Marks DI, Durrant J, McMillan A, Franklin IM, Luger S, Ciobanu N, Rowe JM. In adults with standard-risk acute lymphoblastic leukemia, the greatest benefit is achieved from a matched sibling allogeneic transplantation in first complete remission, and an autologous transplantation is less effective than conventional consolidation/maintenance chemotherapy in all patients: final results of the International ALL Trial (MRC UKALL XII/ECOG E2993). Blood. 2008 Feb 15;111(4):1827-33. doi: 10.1182/blood-2007-10-116582. Epub 2007 Nov 29. PMID 18048644
- [Background] Huguet F, Leguay T, Raffoux E, Thomas X, Beldjord K, Delabesse E, Chevallier P, Buzyn A, Delannoy A, Chalandon Y, Vernant JP, Lafage-Pochitaloff M, Chassevent A, Lheritier V, Macintyre E, Bene MC, Ifrah N, Dombret H. Pediatric-inspired therapy in adults with Philadelphia chromosome-negative acute lymphoblastic leukemia: the GRAALL-2003 study. J Clin Oncol. 2009 Feb 20;27(6):911-8. doi: 10.1200/JCO.2008.18.6916. Epub 2009 Jan 5. PMID 19124805
- [Background] Marks DI, Forman SJ, Blume KG, Perez WS, Weisdorf DJ, Keating A, Gale RP, Cairo MS, Copelan EA, Horan JT, Lazarus HM, Litzow MR, McCarthy PL, Schultz KR, Smith DD, Trigg ME, Zhang MJ, Horowitz MM. A comparison of cyclophosphamide and total body irradiation with etoposide and total body irradiation as conditioning regimens for patients undergoing sibling allografting for acute lymphoblastic leukemia in first or second complete remission. Biol Blood Marrow Transplant. 2006 Apr;12(4):438-53. doi: 10.1016/j.bbmt.2005.12.029. PMID 16545728